CLINICAL TRIAL: NCT01067911
Title: Optimizing Dietary Fatty Acids to Lower Metabolic Risk Factors Among Canadians
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough enrollment, study needs to be revised
Sponsor: University of British Columbia (Other)
Collaborators: Flax Council of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: H09-00188
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Postprandial Lipaemia
Keywords: Postprandial lipids; test meal; fatty acids
MeSH Terms: interventions — Butter; Linseed Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): In this study subjects will consume test meals containing vegetable oils (soy) and butter
  Interventions: Dietary Supplement: Butter and Vegetable oils from soy, flaxseed, high oleic safflower and canola
- 2 (Active Comparator): In this study subjects will consume test meals containing vegetable oils (flaxseed) and butter
  Interventions: Dietary Supplement: In this study subjects will consume test meals containing vegetable oils (soy, flaxseed, high oleic safflower and canola) and butter
- 3 (Active Comparator): In this study subjects will consume test meals containing vegetable oils (high oleic safflower) and butter
  Interventions: Dietary Supplement: In this study subjects will consume test meals containing vegetable oils (soy, flaxseed, high oleic safflower and canola) and butter
- 4 (Active Comparator): In this study subjects will consume test meals containing vegetable oils (canola) and butter
  Interventions: Dietary Supplement: In this study subjects will consume test meals containing vegetable oils (soy, flaxseed, high oleic safflower and canola) and butter

INTERVENTIONS:
Dietary Supplement: Butter and Vegetable oils from soy, flaxseed, high oleic safflower and canola — Test meals prepared with different common fats and oils and consumed by test subjects. Postprandial lipids will be assessed for 6 hours after the consumption of the test meal.
  Arms: 1
Dietary Supplement: In this study subjects will consume test meals containing vegetable oils (soy, flaxseed, high oleic safflower and canola) and butter — Test meals prepared with different common fats and oils and consumed by test subjects. Postprandial lipids will be assessed for 6 hours after the consumption of the test meal.
  Arms: 2
Dietary Supplement: In this study subjects will consume test meals containing vegetable oils (soy, flaxseed, high oleic safflower and canola) and butter — Test meals prepared with different common fats and oils and consumed by test subjects. Postprandial lipids will be assessed for 6 hours after the consumption of the test meal.
  Arms: 3
Dietary Supplement: In this study subjects will consume test meals containing vegetable oils (soy, flaxseed, high oleic safflower and canola) and butter — Test meals prepared with different common fats and oils and consumed by test subjects. Postprandial lipids will be assessed for 6 hours after the consumption of the test meal.
  Arms: 4

SUMMARY:
Scientists believe that what happens to dietary fats after they are eaten, especially how they cleared from the blood, affects risks of heart disease and diabetes is more important than measuring blood fats after an overnight fast. Little is known about what happens in the 6-8 hours after eating common oils available in Canada such as soybean, canola, olive, sunflower or flax oils. Vegetable oils have different types of fatty acids. This study will gather information on what happens to these fatty acids after they are eaten in a meal. The purpose of this research is to show that clearance of fat from the blood varies with the type of vegetable oil in a meal.

DETAILED DESCRIPTION:
The purpose of the present studies is to show that the types of vegetable oil in a meal alter postprandial lipaemia and the transport of n-3 fatty acids. The hypothesis is that a meal which is low in 18:2n-6 and high in the monounsaturated fatty acid 18:1n-9 and 18:3n-3 will result in lower postprandial lipaemia and higher long chain n-3 fatty acids in the unesterified fatty acids when compared to the same meal either high 18:2n-6 and low 18:3n-3. The specific objectives are to determine the magnitude and duration of the increase in plasma TG and the fatty acid composition of chylomicron, LDL and HDL and unesterified fatty acids over 8 hours following the intake of a standard meal with approx 35- 40% energy from fat containing different vegetable oils. The objectives are to show that amount and balance of 18:1n-9, 18:2n-6 and 18:3n-3 in the meal is an important determinant of the extent and duration of postprandial lipaemia, and the appearance of 18:3n-3 and its metabolites in TG and unesterified fatty acids. We will use test meals prepared with different amounts of common fats and oils to provide varying 18:2n-6, 18:3n-3 and 18:1n-9. All the meals will provide less than 10% energy as saturated fatty acids with approx 35% total energy from fat. We also aim to identify the most useful single time point to show differences in plasma post-prandial lipaemia and fatty acids for use in studies in which sequential, repeated blood sampling in the post meal phase is not practical.

Subject characteristics and baseline parameters will be presented using descriptive statistics. Differences in the TG response among subjects and different fats and oils will be assessed using ANOVA, with the use of ANCOVA. Differences in fatty acids at the same time point among the diets will be compared using ANOVA. Prior to analysis, all data will be checked and for those displaying non normal distributions. A P-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, with BMI > 19 < 28 kg/m2
* Waist circumference < 102 cm (40 in) for men and < 88 cm (35 in) for women
* No known chronic disease such as diabetes, heart or thyroid disease or disorder of fat metabolism
* Not taking OTC or prescription medications, not following a vegan or vegetarian diet, not taking fish oil
* Willing to avoid some high fat foods and alcohol for two days, then eat a standardized meal with collection of blood samples over the following 8 hours

Exclusion Criteria:

* No elite athletes or those engaged in vigorous physical activity
* Smokers or those with BMI > 28 or <19
* Waist circumference > 102 cm for men and 88 cm for women
* Known chronic disease such as diabetes or disease involving fat metabolism, the heart or thyroid will be excluded from the study
* Subjects who take any routine prescribed or over-the-counter medications, fatty acids, antioxidant or fish oil, those following a vegan or vegetarian diet, and those who are not willing to abstain from alcoholic beverages and high fat foods for 2 days prior to the test meal and not willing to eat a standardized meal and provide blood samples over the following 8 hours

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Outcome Plasma triglyceride and fatty acids after eating an oil or fat | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Innis, Dr., Principal Investigator — University of British Columbia
Locations (1):
- Child & Family Research Institute, BC Children's Hospital, Vancouver, British Columbia, Canada